CLINICAL TRIAL: NCT05181579
Title: Efficacy of Manual Therapy and Sacroiliac Joint Injection in the Treatment of Patients With Sacroiliac Joint Dysfunction
Brief Title: Efficacy of Manual Therapy and Sacroiliac Joint Injection in Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25
Record Dates: First submitted 2021-12-03; First posted 2022-01-06 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Sacroiliac Joint Somatic Dysfunction
Keywords: Sacroiliac joint dysfunction; Manuel therapy; Sacroiliac joint injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manuel therapy and exercise group (Experimental): Patients in the manual therapy group will receive 5 sessions of sacroiliac joint manipulation once a week. And home exercises will be given and told. Each patient will do exercise 4 days a week for 4 weeks.
  Interventions: Other: Manuel therapy
- Sacroiliac injection and exercise group (Experimental): To patients in the injection group corticosteroid (1 ml 40 mg methylprednisolone) and local anesthetic (1 ml 1% lidocaine)will be injected into the sacroiliac joint using a 22 G spinal needle, guided by fluoroscopy (C-arm fluoroscopy).
  And home exercises will be given and told. Each patient will do exercise 4 days a week for 4 weeks.
  Interventions: Other: Sacroiliac joint injection

INTERVENTIONS:
Other: Manuel therapy — Some sacroiliac manipulation and mobilization techniques will be applied to patients by an experienced physiatrist. Patients in the manual therapy group will receive 5 sessions of sacroiliac joint manipulation once a week.
  Arms: Manuel therapy and exercise group
Other: Sacroiliac joint injection — Corticosteroid (1 ml 40 mg methylprednisolone) and local anesthetic (1 ml 1% lidocaine) will be injected into the sacroiliac joint using a 22 G spinal needle, guided by fluoroscopy (C-arm fluoroscopy) by an experienced physiatrist. It will be applied just one time.
  Arms: Sacroiliac injection and exercise group

SUMMARY:
The purpose of this study is to compare the efficacy of manual therapy and sacroiliac joint injections in patients with sacroiliac joint dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Low back and/or gluteal pain and/or groin pain without radicular extension below the L4 level for more than 3 months
* Pain score greater than 3 according to NRS
* Unresponsiveness to conservative treatment (such as exercise, NSAID)
* At least 3 of the five sacroiliac provocation tests (FABER (Patrick), thigh thrust, Gaenslen, sacroiliac compression, and sacroiliac distraction tests) are positive

Exclusion Criteria:

* Refusing to participate in the study
* Pregnancy
* History of inflammatory disease (ankylosing spondylitis, psoriatic arthritis, rheumatoid arthritis, etc.)
* Infective sacroiliitis
* Malignancy
* Osteoporosis
* Mechanical lumbosacral pathologies (spondylolisthesis, scoliosis, stenosis, etc.)
* Neurological finding in the lower extremity
* Pain spreading below the knee
* History of spinal surgery
* History of allergy to drugs to be injected (local anesthetic, contrast material, steroid allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale, NRS | Change from baseline NRS at 3 months
  NRS is an 11-grade scale that evaluates the severity of pain in adults .NRS is one of the most commonly used scales in the assessment of pain severity. Possible scores ranges from 0( no pain) to 10 ( worst pain)

SECONDARY OUTCOMES:
Oswestry Disability index | Baseline, Month 1, Month 3, Month 6
  The Oswestry disability index will be used to evaluate how much the patients' low back pain limits their activities in daily life. This index was first created in 1980 . The questionnaire consists of 10 sections, each assessing limitations in different daily activities and functions. Each section is scored from 0 to 5. A score of 0 indicates that there is no restriction while doing that activity, while a score of 5 represents the highest level of restriction in that activity. The maximum score is 50. As the total score increases, the disability level of the individual increases. In 2004, Turkish validity study was carried out by Yakut et al.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Guzelkucuk, MD, Study Director — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No